CLINICAL TRIAL: NCT02159105
Title: Abdominal Ultrasound Assessment in the Post-cesarean Patient
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dana Gossett, Assistant Professor, Northwestern University
Other Study IDs: STU00080804
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Postpartum Hemorrhage; Postsurgical Bleeding; Abdominal Ultrasound; FAST Scan; Non-invasive Hemoglobin Measurement
Keywords: postpartum hemorrhage; postsurgical bleeding; abdominal ultrasound; FAST scan; non-invasive hemoglobin measurement
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing cesarean delivery: FAST scan and non-invasive hemoglobin measurement
  Women undergoing cesarean delivery will undergo a non-invasive hemoglobin measurement both before and after surgery. An abdominal ultrasound will be performed to establish normal levels of intra-abdominal fluid after cesarean delivery.
  Interventions: Device: FAST scan and non-invasive hemoglobin measurement

INTERVENTIONS:
Device: FAST scan and non-invasive hemoglobin measurement — A "FAST scan", or abdominal ultrasound will be performed within one hour of cesarean delivery to establish normal levels of postoperative intraabdominal fluid.
  Women will also have their hemoglobin measured via a non-invasive method, the Masimo Pronto 7, at 3 time points: immediately prior to surgery (within 2 hours), immediately after surgery (within 1 hour), and the morning following surgery (within 24 hours).
  Other Names: Masimo Pronto 7; FAST scan

SUMMARY:
This study is designed to see if abdominal ultrasound after planned cesarean delivery can identify women with ongoing intra-abdominal bleeding.

DETAILED DESCRIPTION:
Hemorrhage is the second leading cause of maternal mortality in the United States. Women have an increased risk of hemorrhage after cesarean sections.Uterine atony is the culprit in 80% of cases, but in the post-operative patient, an intra-abdominal bleed requiring a return to the operating room must also be considered. The Focused Assessment with Sonography in Trauma (FAST) has been used in the emergency department to evaluate for intra-abdominal bleeding after trauma. FAST evaluation has not been studied in the post-operative period for evaluation for intra-abdominal bleeding. Ultrasound is a rapid and readily-available modality for this type of evaluation, and obstetricians are already familiar with the technology. But one must be cautious, as a certain amount of free fluid on CT is common in the postoperative patient. Before basing clinical decisions on a FAST scan, we much determine how much fluid is normal in a patient after cesarean delivery. We hypothesize that a certain amount of fluid in the abdomen visualized by ultrasound may be normal after a cesarean delivery, and that for ultrasound to become a valuable modality to assess for intra-abdominal bleeding in the post-cesarean patient, the amount of normal fluid must be determined. However, in order to interpret what an "appropriate" amount of fluid would be, we will also need an assessment of patient hemoglobin levels. Thus, we would additionally plan to validate a rapid, non-invasive hemoglobin measurement for use in the post-cesarean obstetric patient. The Pronto7 device measures the blood's absorption of multiple wavelengths of light to determine hemoglobin. The device avoids a blood draw and its associated pain. It also provides immediate results. We anticipate that we will identify an association between the amount of fluid seen on ultrasonographic evaluation after cesarean delivery and adverse outcomes such as larger than expected decrease in hemoglobin, need for transfusion and need for take-back to the operating room. We also anticipate that the use of non-invasive hemoglobin measurements may provide a rapid, painless assessment of postoperative hemoglobin; this may allow us to identify patients who merit earlier postoperative monitoring with a traditional CBC. It may also allow us to identify women who do not need an invasive CBC on postoperative day 1, which may decrease blood draws and costs in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 18 years of age or older
* English-speaking
* Non-urgent cesarean sections

Exclusion Criteria:

* Preeclampsia/eclampsia
* <18 years old
* Urgent/emergent cesarean section
* Not English-speaking
* Unable to consent

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women undergoing non-emergent cesarean delivery at Prentice Women's Hospital, who speak English and are able to provide consent, will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
FAST Scan results | 1 hour
  Abdominal ultrasound will be performed within 1 hour of surgery completion. Studies will be classified as positive or negative, and the amount and location of intra-abdominal fluid will also be documented.

SECONDARY OUTCOMES:
Non-invasive hemoglobin measurement | 1 day
  Non-invasive hemoglobin measurements will be taken immediately prior to surgery (baseline measurement), immediately postoperatively, and on the morning of postoperative day 1 (within 24 hours of surgery). The results of the final measurement will be compared to the standard blood draw on postoperative day one of a routine complete blood count (CBC) to assess the accuracy of this non-invasive measurement technique among postpartum women.

CONTACTS AND LOCATIONS:
Overall Officials: Dana R Gossett, MD, MSCI, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Hoppenot C, Tankou J, Stair S, Gossett DR. Sonographic evaluation for intra-abdominal hemorrhage after cesarean delivery. J Clin Ultrasound. 2016 May;44(4):240-4. doi: 10.1002/jcu.22289. Epub 2015 Aug 24. PMID 26302357